CLINICAL TRIAL: NCT00793338
Title: Evaluation of Sildenafil for the Treatment of Moderate Congestive Heart Failure
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The project was not funded and could not be initiated.
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Joe R. Anderson, Associate Professor of Pharmacy Practice and Administrative Sciences, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRRC 05-369
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
Keywords: Heart failure; Sildenafil; Cardiopulmonary exercise test; quality of life; 6 minute walk test
MeSH Terms: conditions — Heart Failure | interventions — Sildenafil Citrate; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sildenafil (Experimental): All patients will receive open-label treatment with sildenafil.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Sildenafil 20mg three times a day for 3 months.
  Other Names: Heart failure; Cardiopulmonary exercise test

SUMMARY:
The purpose of the study is to evaluate whether sildenafil helps treat heart failure. Some patients with heart failure have high blood pressure in the lungs (referred to as "pulmonary hypertension"). Sildenafil is a medication that is used to treat high blood pressure in the lungs and may reduce symptoms of heart failure. Studies have looked at the short-term benefit of sildenafil in patients with congestive heart failure, but this study will look at the longer-term benefits of 12 weeks of therapy with sildenafil.

DETAILED DESCRIPTION:
Objective: To determine the effect of acute and long-term treatment with sildenafil on the clinical status of patients with moderate HF. Secondary Objectives: To determine the effect of acute and long-term treatment with sildenafil on cardiopulmonary exercise performance, the effect of acute and long-term treatment with sildenafil on neurohormonal activation, the effect of acute and long-term treatment with sildenafil on hemodynamics, and the effect of long-term treatment with sildenafil on quality of life. Background: Secondary pulmonary hypertension (PH) is a frequent manifestation of heart failure resulting in impaired vascular reactivity and permeability which contributes to the symptoms of HF. Levels of endothelin-1 (ET-1), a potent vasoconstrictor, are increased in patients with HF. At the same time, pulmonary artery nitric oxide (NO) production is decreased. NO increases concentrations of the second messenger cyclic-GMP, ultimately leading to vasodilation. This imbalance between NO-dependent vasodilation and ET-1 induced vasoconstriction likely contributes to the development of secondary pulmonary hypertension. cGMP is metabolized by the type 5 isoform of phosphodiesterase (PDE5) an enzyme that is highly expressed in the lung. Sildenafil, a selective PDE5 inhibitor, has been used extensively for the treatment of erectile dysfunction and has recently been approved for use in the treatment of PH. Recent studies of short-term administration of sildenafil in HF patients with secondary PH have demonstrated reductions in pulmonary arterial pressure, pulmonary vascular resistance, pulmonary capillary wedge pressure, and systemic vascular resistance while increasing cardiac index and exercise performance. However, it remains to be seen if sildenafil is safe and effective in the long-term treatment of heart failure. Methods: This will be an open-label, pilot study designed to evaluate the safety and efficacy of sildenafil for the treatment of moderate heart failure. The primary endpoint will be change in 6-minute walk test distance. Secondary endpoints will be changes in peak oxygen consumption (measured by cardiopulmonary exercise testing), neurohormones (b-type natriuretic peptide, catecholamines, ET-1), quality of life scores. Additionally, we will attempt to analyze responsiveness to sildenafil on the basis of PDE5 polymorphisms. Study procedures will be performed at the UNM General Clinical Research Center and the UNM Congestive Heart Failure Clinic. Patients will be hospitalized for 3 days to analyze safety and efficacy of sildenafil administered three times daily. Patients will complete exercise testing, neurohormone, and hemodynamic assessments at baseline (day 1) and following 24 hours of sildenafil treatment. The patients will then be discharged to complete a 12-week maintenance phase of treatment. At the conclusion of the maintenance phase the patients will be readmitted for 2 day to have repeat measurements performed. The main analysis will be done using paired t-tests. All statistical analysis will be performed using SAS v6.12.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Diagnosis of chronic heart failure with an ejection fraction less than or equal to 45% per either an echocardiogram, nuclear cardiolyte stress test, or cardiac catheterization performed within the past 6 months.
* New York Heart Association Functional Class III
* Must be on optimal heart failure therapy according to AHA/ACC heart failure guidelines, including treatment with ACEI and beta-blocker therapy, or have documented rationale for variation, including intolerance, contraindication, patient preference, or personal physician's judgment

Exclusion Criteria:

* Comorbid disease or behavioral or other limitations that: 1) interfere with performing exercise test, or 2) prevent completion of 12 week study
* Currently pregnant or intent to become pregnant in the next 12 weeks or currently breastfeeding.
* Major cardiovascular event or cardiovascular procedure within the prior 6 weeks
* History of Chronic Obstructive Pulmonary Disease or Reactive Airway Disease
* Known hypersensitivity to sildenafil
* Current use of medications known to be a potent inhibitor of CYP3A4 (e.g., ritonavir, ketoconazole, itraconazole)
* Current or recent (within 6 months) use of organic nitrate medications (e.g. isosorbide dinitrate, sublingual nitroglycerin)
* Known diagnosis of pulmonary veno-occlusive disease or non-arteritic anterior ischemic optic neuropathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Change in 6-minute walk distance | 24 hours and 3 months

SECONDARY OUTCOMES:
Changes in peak oxygen consumption (measured by cardiopulmonary exercise testing) | 24 hours and 3 months
Change in the level of neurohormones (b-type natriuretic peptide, catecholamines, ET-1), | 24 hours and 3 months
Change in quality of life | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Joe R Anderson, PharmD, Principal Investigator — University of New Mexico College of Pharmacy
Locations (1):
- Clinical Translational Science Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided